CLINICAL TRIAL: NCT06675877
Title: Impact of Virtual Reality on Pain, Anxiety and Depression in Pediatric Patients with ESRD on Regular Hemodialysis Through Arteriovenous Fistula.
Brief Title: Impact of Virtual Reality on Pediatric Patients with ESRD on Regular Hemodialysis Through Arteriovenous Fistula.
Acronym: VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, lecturer of pediatrics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VR on HD children
Record Dates: First submitted 2024-10-22; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Pain; Anxiety
Keywords: VR; pediatric
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: the child lay on the bed and wore virtual reality eyeglasses, the eyeglasses were placed on the child's head, the child watched 3 D VR kids' cartoons or videos to distract his/her attention during needle insertion. The video was displayed through a smart phone inserted inside the virtual reality headset.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): Group A Cases only will receive in each dialysis session standard care together with VR camera.
  Interventions: Other: virtual reality camera
- group B (No Intervention): Group B control group undergo three to four dialysis sessions weekly; they will receive the standard care only in their dialysis sessions without VR camera

INTERVENTIONS:
Other: virtual reality camera — The virtual reality eyeglasses were placed on the child's head, the child watched 3 D VR kids' cartoons or videos to distract his/her attention during needle insertion. The video was displayed through a smart phone inserted inside the virtual reality headset.
  Arms: group A

SUMMARY:
This case control study will be conducted to study the effectiveness of Virtual Reality technique on pain during arteriovenous cannulation and on reduction of anxiety and depression in Pediatric Patients with ESRD undergoing regular hemodialysis through arteriovenous fistula.

DETAILED DESCRIPTION:
This case control study will be conducted at nephrology and dialysis Unit Pediatric Department Tanta University Hospital (TUH) for a period of 6 months starting from April 2024.This study will be conducted on convenient sample of 60 participants. they will be classified as follow group A (cases) Group B (controls)each group will contain 30 children and adolescents with end stage renal disease on regular hemodialysis for three times weekly at our nephrology Unit at TUH during the period of the study

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with end stage renal disease aged from 8 to 18 years on regular hemodialysis through functioning arteriovenous fistula and are fully oriented with time, persons and place at time of data collection. All participants either cases or controls suffer from anxiety, depression or both.

Exclusion Criteria:

* Children with temporary or permanent catheter for dialysis.
* Children with mental illness, visual and auditory defects.
* Children took any pharmacological pain reliever or antipsychotic drugs.
* Non anxious or depressed Children.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
SCARED for anxiety Screen for Child Anxiety Disoders {SCARED} Child, parent version: It is a self-report screening questionnaire for anxiety disorders during hemodialysis | 6 months
  The SCARED is useful for generalized anxiety disorder, social anxiety disorder, phobic disorders, and potentially school anxiety problems. Cases and controls will be asked to complete the questionnaire before entering the study (examination No. I) and after its completion after 3 months (examination No. II).

SECONDARY OUTCOMES:
The Children's Depression Inventory scale for depression during hemodialysis | 6 months
  Cases and controls will be asked to complete the questionnaire of The Children's Depression Inventory scale before entering the study (examination No. I) and after its completion after 3 months (examination No. II).

CONTACTS AND LOCATIONS:
Overall Officials: sara Ma ElGhoul, MD, Principal Investigator — Tanta university hospital
Locations (1):
- Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
for confidence